CLINICAL TRIAL: NCT02021630
Title: The Collateral Impact of Bariatric Surgery on Families
Acronym: Collateral
Status: Completed | Type: Observational
Sponsor: Geisinger Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 2012-0360; SRC-L-15 (Registry Identifier: Geisinger's Scientific Review Committee)
Record Dates: First submitted 2013-12-20; First posted 2013-12-27 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-07

CONDITIONS: Obesity; Bariatric Surgery Candidate; Weight Loss
Keywords: Obesity; Bariatric Surgery; Weight Loss; Physical Activity; Body Composition
MeSH Terms: conditions — Obesity; Weight Loss; Motor Activity | interventions — Treatment Outcome

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Patient: No intervention will occur during this study. Evaluation of changes in patients' family after having patient has bariatric surgery.
  Interventions: Other: Outcomes
- Spouse/Partner: No intervention will occur during this study. Evaluation of changes in patients' family after having patient has bariatric surgery.
  Interventions: Other: Outcomes
- Child(ren): No intervention will occur during this study. Evaluation of changes in patients' family after having patient has bariatric surgery.
  Interventions: Other: Outcomes

INTERVENTIONS:
Other: Outcomes — No intervention will occur during this study. Evaluation of changes in patients' family after having patient has bariatric surgery.

SUMMARY:
This proposal is designed to examine the impact of bariatric surgery on the health of patients and their families. The shared environment of spouses/cohabitating partners suggests that patients' families are exposed to the extensive diet and lifestyle changes required of patients following bariatric surgery.

DETAILED DESCRIPTION:
The specific aims of this proposal are to:

1. Collect clinical data (e.g., weight, blood pressure, body composition, blood sample), as well as monitor physical activity and eating patterns, before and after bariatric surgery (Adults Only).
2. Analyze clinical data, physical activity and eating patterns to determine how the health of patients and their families change after one family member completes bariatric surgery (Adults Only).
3. Determine the feasibility of recruiting patients, spouses/partners and their children.

ELIGIBILITY:
Inclusion Criteria:

* All patients who receive surgery have been cleared medically and psychosocially for surgery. Thus, surgical candidacy criteria will serve as eligibility criteria for the current study for surgical patients.
* Cohabitation with patients will be considered inclusion criteria for partners/spouses.
* Children between the ages of ≥5 - ≤ 16, who cohabitate with the patient the majority of the time will be asked to participate by providing assent.

Exclusion Criteria:

* Report current or planned use of weight loss medications (including OTC), or other weight loss strategy.
* Report pregnancy, lactation, or plans to become pregnant during study duration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients enrolled in the bariatric surgery program at Geisinger Medical Center's Center for Nutrition and Weight Management along with their spouse/partner and/or child(ren) ages 5-16.
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2012-12; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Weight | Pre-operatively, post-operatively 6 months and 12 months

SECONDARY OUTCOMES:
Percent body fat | Pre-operatively, post-operatively 6 months and 12 months
Physical Activity | Pre-operatively, post-operatively 6 months and 12 months
  Accelerometer

OTHER OUTCOMES:
Laboratory outcomes | Pre-operatively, post-operatively 6 months and 12 months
  Lipid panel, insulin, glucose
Questionnaires | Pre-operatively, post-operatively 6 months and 12 months
  Home Food Inventory, Social Support

CONTACTS AND LOCATIONS:
Overall Officials: Christopher D Still, DO, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger Clinic, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided